CLINICAL TRIAL: NCT00002531
Title: MULTICENTRE TRIAL OF INTENSIFIED THERAPY FOR ADULT ALL (O5/93)
Brief Title: Combination Chemotherapy in Treating Adults With Acute Lymphocytic Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000078421; GER-GMALL-ALL-05/93; EU-93002
Record Dates: First submitted 1999-11-01; First posted 2004-02-16 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2006-12

CONDITIONS: Leukemia
Keywords: untreated adult acute lymphoblastic leukemia; T-cell adult acute lymphoblastic leukemia; B-cell adult acute lymphoblastic leukemia; non-T, non-B adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Doxorubicin; Etoposide; Ifosfamide; Leucovorin; Mercaptopurine; Methotrexate; Mitoxantrone; Prednisolone; Teniposide; Thioguanine; Vincristine; Vindesine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Drug: asparaginase
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: leucovorin calcium
Drug: mercaptopurine
Drug: methotrexate
Drug: mitoxantrone hydrochloride
Drug: prednisolone
Drug: teniposide
Drug: thioguanine
Drug: vincristine sulfate
Drug: vindesine
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Randomized phase II trial to study the effectiveness of various combination chemotherapy regimens in treating patients with acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Develop risk-adapted therapy for patients with low-risk, high-risk, T-cell, or B-cell acute lymphocytic leukemia (ALL). II. Determine the complete remission rate in these patients treated with the following strategies: increased doses of cyclophosphamide during induction and reinduction, early use of high-dose cytarabine plus mitoxantrone (for high-risk patients), and increased doses of methotrexate (for B-cell ALL patients). III. Determine the duration of remission and survival of patients in all risk groups treated with intensified consolidation and subtype-specific chemotherapy. IV. Compare the effects of intensified vs conventional maintenance therapy in patients of all risk groups.

OUTLINE: This is a randomized, multicenter study. Patients are assigned to 1 of 4 treatment groups based on disease status. Patients in groups 1-3 with a large leukemic cell mass, in particular those with a WBC greater than 25,000/mm3 and/or marked organomegaly, receive preinduction therapy comprising oral prednisolone (PRDL) 3 times a day on days 1-7 and vincristine (VCR) IV on day 1. Group 1 (low-risk acute lymphocytic leukemia (ALL)): First induction therapy: Patients receive oral PRDL 3 times a day on days 1-7 of weeks 1-4, asparaginase (ASP) IV over 30 minutes on days 1-7 of weeks 3 and 4, VCR IV and daunorubicin IV over 30 minutes on day 1 of weeks 1-4, and methotrexate (MTX) IT on day 1 of week 1. Patients who achieve complete remission (CR) after first induction therapy proceed to first consolidation therapy on group 1. Second induction therapy: Patients receive oral cyclophosphamide (CTX) IV on day 1 of weeks 5, 7, and 9; cytarabine (ARA-C) IV over 1 hour or subcutaneously on days 3-6 and MTX IT on day 3 of weeks 5-8; and oral mercaptopurine (MP) on days 1-7 of weeks 5-8 and day 1 of week 9. Patients who achieve CR during second induction therapy undergo prophylactic cranial irradiation 5 days a week for 2.4 weeks. Patients who achieve CR after second induction therapy proceed to group 3. First consolidation therapy: Patients receive high-dose MTX IV continuously with leucovorin calcium (CF) rescue on day 1, ASP IV over 1 hour on day 2, and oral MP on days 1-5 of weeks 13 and 15; and teniposide (VM-26) IV over 1 hour and ARA-C IV over 1 hour on days 1-5 of week 17. Triple intrathecal therapy (TIT) comprising MTX, ARA-C, and dexamethasone (DM) is also administered on day 1 of week 17. First reinduction therapy: Patients receive oral PRDL three times a day on days 1-7 and VCR IV and doxorubicin (DOX) IV over 30 minutes on day 1 of weeks 21-24, and TIT on day 1 of week 21. Second reinduction therapy: Patients receive CTX IV and TIT on day 1 of week 25, and ARA-C IV over 1 hour on days 3-6 and oral thioguanine (TG) on days 1-7 of weeks 25 and 26. Second consolidation therapy: Patients receive oral MP daily and oral MTX weekly during weeks 29-32, 34-38, 40-44, 46-50, and 52; high-dose MTX, CF rescue, and ASP as in first consolidation therapy during weeks 33 and 45; and VM-26, ARA-C, and TIT as in first consolidation therapy during weeks 39 and 51. Group 2 (T-cell ALL with or without mediastinal involvement): First induction therapy: Patients receive treatment as in first induction therapy on group 1. Patients with residual tumor greater than 2 cm after first induction therapy also undergo mediastinal radiotherapy 5 days a weeks for 2.4-2.7 weeks concurrently with prophylactic cranial irradiation. Second induction therapy: Patients receive treatment as in second induction therapy on group 1. First consolidation therapy: Patients receive high-dose ARA-C IV over 3 hours every 12 hours on days 1-4 and mitoxantrone (DHAD) IV over 30 minutes on days 3-5 during week 13; and high-dose MTX, CF rescue, ASP, and MP as in first consolidation therapy on group 1 during week 17. First reinduction therapy: Patients receive treatment as in first reinduction therapy on group 1. Second reinduction therapy: Patients receive treatment as in second reinduction therapy on group 1. Second consolidation therapy: Patients receive MP and MTX as in second consolidation therapy on group 1; CTX IV, ARA-C IV continuously, and TIT on day 1 during weeks 33 and 45; and VM-26, ARA-C, and TIT as in first consolidation therapy on group 1 during weeks 39 and 51. Group 3 (high-risk ALL): First induction therapy: Patients receive treatment as in first induction therapy on group 1. Second induction therapy: Patients receive CNS-effective chemotherapy comprising high-dose ARA-C every 12 hours on days 1-4 and DHAD IV over 30 minutes on days 3-5 during week 6. First consolidation therapy: Patients receive high-dose MTX, CF rescue, and ASP as in first consolidation therapy on group 1; and CTX, ARA-C, and TIT as in second consolidation therapy on group 2 during week 17. First reinduction therapy: Patients receive treatment as in first reinduction therapy on group 1. Second reinduction therapy: Patients receive treatment as in second reinduction therapy on group 1. Second consolidation therapy: Patients receive MP and MTX as in second consolidation therapy on group 1; treatment as in second induction therapy on group 3 during week 33; high-dose MTX, CF rescue, ASP, and MP as in first consolidation therapy on group 1 during week 39; CTX, ARA-C, and TIT as in second consolidation therapy on group 2 during week 45; and VM-26, ARA-C, and TIT as in first consolidation therapy on group 1 during week 51. Groups 1-3: Patients who are age 15 to 50, achieve first CR, and have a suitable donor undergo allogeneic bone marrow transplantation. Patients who are under age 40 undergo bone marrow transplantation from a matched unrelated donor. Patients who have Philadelphia chromosome/bcr-abl positive disease and no suitable donor undergo purged autologous peripheral blood stem cell transplantation instead of reinduction therapy during first CR. CNS therapy: Patients with CNS disease at entry receive TIT 2 or 3 times weekly beginning immediately upon diagnosis and continuing until 5 doses after blasts are cleared from the CSF. Patients on group 1 and 2 undergo irradiation of the entire neuraxis 5 days a week for 2.7-3.2 weeks during second induction therapy. Maintenance therapy: After completion of 1 year of treatment on group 1, 2, or 3, patients are randomized to 1 of 2 treatment arms. Arm I: Patients receive MP daily and MTX weekly on odd-numbered months between months 13-30; CTX, ARA-C, and TIT as in second consolidation therapy on group 2 during months 14, 20, and 26; VM-26, ARA-C, and TIT as in first consolidation therapy on group 1 during months 16, 22, and 28; and high-dose MTX, CF rescue, and ASP as in first consolidation therapy on group 1 during months 18, 24, and 30. Arm II: Patients receive MP plus MTX as in second consolidation therapy on group 1 continuously and TIT every 2 months during months 13-30. Group 4 (B-cell ALL): Pretreatment: Patients who are age 50 and under receive CTX IV over 1 hour and oral PRDL 3 times a day on days 1-5. Patients who are over age 50 receive CTX IV and oral DM on days 1, 3, and 5. Treatment: Patients receive alternating therapy on blocks A and B. Block A therapy consists of VCR IV, MTX IV continuously, and CF rescue on day 1; ifosfamide IV over 1 hour and oral DM on days 1-5; VM-26 IV over 1 hour and ARA-C IV over 1 hour every 12 hours on days 4 and 5; and TIT on days 1 and 5. Block B therapy consists of VCR IV, MTX IV continuously, and CF rescue on day 1; CTX IV over 1 hour and oral DM on days 1-5; DOX IV over 15 minutes on days 4 and 5; and TIT on days 1 and 5. Blocks A and B continue every 3 weeks for a total of 6 courses. Patients who have not achieved CR after 3 courses or who develop disease progression at any time may optionally receive vindesine, ARA-C, etoposide, and DM. Patients with CNS disease undergo craniospinal irradiation after 2 courses of systemic chemotherapy (block A and B therapy). Patients receive TIT 2-3 times weekly until CSF is clear after block A therapy only if response is unsatisfactory.

PROJECTED ACCRUAL: Approximately 700 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of low-risk acute lymphocytic leukemia (ALL) (common ALL or pre-B-cell) Must meet 1 of the following 2 conditions: Age 51 to 65 and meets the following criteria: No mediastinal mass No T-cell or B-cell disease Age 15 to 50 and meets the following criteria: Philadelphia chromosome (Ph) negative bcr-abl negative Initial WBC less than 30,000/mm3 OR Diagnosis of T-cell ALL with or without mediastinal involvement Age 15 to 50 OR Diagnosis of high-risk ALL (common ALL or pre-B-cell) Age 15 to 50 and meets 1 of the following criteria: Ph positive bcr-abl positive Pre-pre-B-cell disease, i.e., t(4;11) Initial WBC greater than 30,000/mm3 OR Diagnosis of B-cell ALL

PATIENT CHARACTERISTICS: Age: See Disease Characteristics 15 to 65 Performance status: Not specified Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Not specified Renal: No renal failure Cardiovascular: No cardiomyopathy Other: HIV-1 and HIV-2 negative No severe psychiatric disease

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior cytostatic drugs except vincristine Endocrine therapy: Prior corticosteroids allowed Radiotherapy: Not specified Surgery: Not specified Other: No more than 2 weeks of prior therapy No other prior cytostatic drugs

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-01

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hoelzer, MD, PhD, Study Chair — Johann Wolfgang Goethe University Hospital
Locations (1):
- Klinikum der J.W. Goethe Universitaet, Frankfurt, Germany

REFERENCES:
- [Background] Bruggemann M, Raff T, Flohr T, Gokbuget N, Nakao M, Droese J, Luschen S, Pott C, Ritgen M, Scheuring U, Horst HA, Thiel E, Hoelzer D, Bartram CR, Kneba M; German Multicenter Study Group for Adult Acute Lymphoblastic Leukemia. Clinical significance of minimal residual disease quantification in adult patients with standard-risk acute lymphoblastic leukemia. Blood. 2006 Feb 1;107(3):1116-23. doi: 10.1182/blood-2005-07-2708. Epub 2005 Sep 29. PMID 16195338
- [Background] Burmeister T, Goekbuget N, Schwartz S, et al.: Outcome of adult ALL patients with fusion transcript E2A-PBX1: results from the GMALL therapy trials 5/93 and 6/99. [Abstract] Blood 108 (11): A-1888, 2006.